CLINICAL TRIAL: NCT05496634
Title: Investigation of Biopsychosocial Characteristics of Individuals Doing Pilates and Sedentary Individuals During the Covid-19 Pandemic Process
Brief Title: The Effect of Pilates on Biopsychosocial Characteristics in the Covid-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal Investigator, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-840
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: COVID-19; Healthy; Sedentary; Exercise; Pilates
MeSH Terms: conditions — COVID-19; Sedentary Behavior; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): An informative presentation will be made emphasizing the importance of physical activity during the pandemic process. Individuals in the exercise group also participated in pilates sessions that lasted 50 minutes, 2 days a week for 8 weeks.
  Interventions: Behavioral: Exercise therapy
- Control Group (Experimental): An informative presentation will be made emphasizing the importance of physical activity during the pandemic process.
  Interventions: Behavioral: Sedantary

INTERVENTIONS:
Behavioral: Sedantary — An informative presentation
  Arms: Control Group
Behavioral: Exercise therapy — Pilates exercise therapy
  Arms: Exercise Group

SUMMARY:
The aim of this study is to investigation of biopsychosocial characteristics of individuals who do pilates and sedentary individuals during the COVID-19 pandemic. The study was carried out with 2 groups: individuals ages 20-50,participating in a pilates program for 8 weeks (n:27) and sedentary individuals (n:27). Before starting this study, the groups were assessed for biopsychosocial status with the Cognitive Exercise Therapy Approach- Biopsychosocial Questionnaire (CETA-BQ) , for depression levels with the Beck Depression Inventory (BDI), for covid-19 fear levels with the Coronavirus Anxiety Scale, for their sleep quality with the Pittsburg Sleep Quality Index (PSQI), quality of life was assessed with the Nottingham Health Profile (NHP). After the first evaluation, an informative presentation emphasizing the importance of physical activity during the pandemic process was given to all participants. Individuals in the exercise group also participated in pilates sessions that lasted 50 minutes, 2 days a week for 8 weeks. At the end of 8 weeks, all questionnaires were repeated for both groups.

DETAILED DESCRIPTION:
Coronavirus disease-2019 (COVID-19); It is an infection that emerged in China in December 2019 and then turned into a pandemic, and it still continues to be seen all over the world. After the first case was seen in our country, the government took measures to slow down the coronavirus epidemic and protect the health of the society. While these measures physically affect people's lives, they limited people's range of motion and reduced their physical activity levels. In early March 2020, researchers predicted that social distancing, along with school closures and restrictions, could result in less physical activity, prolonged sedentary behavior, and poor sleep quality. In a study comparing physical activity behaviors before and during isolation as a result of COVID-19, it was shown that COVID-19 isolations cause a negative effect on all physical activity levels and cause more than 28% increase in daily sitting times.

In addition to the physical effects of the coronavirus, there are also psychological effects. Its psychological effects are not limited to individuals infected with the virus, but are also seen in individuals who are not infected. The COVID-19 epidemic, which is accepted as a stress factor, is associated with the concept of death in most individuals due to the disease, the fear of being infected with the virus and the tendency to take extra precautions, the anxiety of transmitting the virus to others, the fear of death, the state of irritability, attention and concentration disorder. Reactions such as fatigue, sleep disturbance, conflict with family members and social withdrawal are also observed. Deterioration of sleep quality facilitates the spread of infectious diseases and negatively affects the mental health and quality of life of individuals. In addition, the frequent pronunciation of the words social distance, isolation and contact in the society has led to the emergence of a new fear, which is expressed in different terms such as "coronaphobia" or "fear of COVID-19".

Physically active individuals generally experience less stress, depression, and anxiety. Studies show that physical activity strengthens the immune system by increasing the number of immune cells in our body. Exercises that can be applied everywhere, such as walking at home, walking to the market by taking protective measures against the disease, sitting on a chair, climbing stairs, pilates and yoga can be counted as examples of the types of exercises that can be done during quarantine periods.

The Pilates exercise method was created by Joseph Pilates in the 1920s and its original name is "Contrology". Pilates method; It is an exercise system that has the principles of concentration, centering, control, precision in movements, movement flow and breathing dynamics (11). Exercises; It is made on a mat or with special equipment with adjustable spring resistance (12). During the First World War, Joseph Pilates began experimenting with spring mattresses to help treat the war-wounded and attached springs to the ends of mattresses to allow patients to exercise against resistance while tied to the bed. He noticed that exercises with resistance improved muscle tone in patients faster than exercises without resistance. As a result, Joseph Pilates developed the Universal Reformer, a sliding platform with springs on which one can sit, lean or stand, and the Cadillac, a mattress with springs on all four sides (13).

No study has been found in the literature examining the biopsychosocial characteristics of pilates and sedentary individuals during the COVID-19 pandemic. In this context, in our study; The biopsychosocial characteristics of individuals doing pilates and sedentary individuals during the COVID-19 pandemic were examined.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-50, without any known neurological, mental, vestibular or orthopedic disease,
* For the exercise group, doing reformer pilates 2 days a week for 8 weeks,
* For the control group, who is not involved in any physical activity in their daily life (sedentary),
* Individuals with at least 2 doses of covid-19 vaccine

Exclusion Criteria:

* Having orthopedic, neurological or musculoskeletal system problems that prevent him from doing reformer pilates,
* Not attending the sessions regularly,
* Pregnancy status or suspected,
* Covid-19 positive participants

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach- Biopsychosocial Questionnaire (CETA-BQ) | 0-8 weeks
  It was used to evaluate the biopsychosocial status of the participants. Each item is scored between 0-4 according to the Likert system. An increase in the score indicates a worsening of the biopsychosocial status. (4: Yes always, 3: Yes often, 2: Yes sometimes, 1: Yes rarely, 0: No, never)
Beck Depression Inventory (BDI) | 0-8 weeks
  Beck Depression Scale consists of 21 items including depressive symptoms. Minimal depression from 0 to 9 points; 10-16 points mild depression; 17-29 points indicate moderate depression and 30-63 points indicate severe depression.
Coronavirus Anxiety Scale | 0-8 weeks
  The scale was created by evaluating the scales evaluating different fear parameters by experts and taking into account the opinions of the participants. The scale is scored in a one-factor and five-point Likert type (1=I strongly disagree; 5=I strongly agree). The scale consists of seven items. The score that can be obtained from the scale is between 7-35. A high score indicates greater fear of COVID-19.
Pittsburg Sleep Quality Index (PSQI) | 0-8 weeks
  The PSQI consists of 7 components: 1. subjective sleep quality, 2. sleep latency, 3. sleep duration, 4. habitual sleep efficiency, 5. sleep disturbance, 6. sleep medication use, 7. daytime dysfunction. Each component is evaluated with a score between 0-3. The total score is between 0-21. A higher score indicates worsening sleep quality. A score of 0-4 is considered good sleep quality, while a score of 5-21 is defined as poor sleep quality.
Nottingham Health Profile (NHP) | 0-8 weeks
  Questionnaire; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items) and emotional reaction (9 items). There are 38 questions in total. Questions are answered with yes or no. Each section is scored between 0-100. Zero indicates best health, 100 indicates worst health.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)